CLINICAL TRIAL: NCT01750346
Title: Placebo Controlled Double Blind Study of Acetyl Hexapeptide-8 in Treatment of Blepharospasm
Brief Title: Acetyl Hexapeptide-8 for Blepharospasm
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 130022; 13-N-0022
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Results first posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-09

CONDITIONS: Focal Dystonia
Keywords: Blepharospasm; Treatment; Dystonia; Acetyl-Hexapeptide
MeSH Terms: conditions — Dystonic Disorders; Blepharospasm; Dystonia | interventions — acetyl-glutamyl-glutamyl-methionyl-glutaminyl-arginyl-argininamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 0.05% AH-8 (Active Comparator): Participants in the 0.05% AH-8 arm received the higher dose of the study drug, Acetyl Hexapeptide 8 (AH-8), which is sold under the brand name, Argireline.
  Interventions: Drug: Topical acetyl hexapeptide-8
- 0.025% AH-8 (Active Comparator): Participants in the 0.025% AH-8 arm received the lower dose of the study drug, Acetyl Hexapeptide 8 (AH-8), which is sold under the brand name, Argireline.
  Interventions: Drug: Topical acetyl hexapeptide-8
- Placebo (Placebo Comparator): Participants in the Placebo arm received the placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical acetyl hexapeptide-8
  Arms: 0.025% AH-8; 0.05% AH-8
Drug: Placebo
  Arms: Placebo

SUMMARY:
Background:

- Blepharospasm is caused by excessive contraction of the muscles that close the eye. One treatment is botulinum neurotoxin (BoNT), which works by weakening those muscles. Like BoNT, acetyl hexapeptide-8 (AH-8) works to weaken the muscles, but is available as a skin cream. AH-8 is the active ingredient in a number of cosmetic creams used to treat wrinkles. Researchers thought that AH-8 cream could be used to treat blepharospasm, but the original dose studied was not very effective. They want to try a higher dose of AH-8 in a cream to see if it can be a more effective treatment.

Objectives:

- To see if AH-8 cream can improve the symptoms of blepharospasm.

Eligibility:

- Individuals at least 18 years of age who have blepharospasm that is severe enough to require treatment.

Design:

* This study will involve up to eight study visits.
* Participants will be screened with a physical exam and medical history. They will answer questions about their symptoms. They will also have a blink test to see how severe the blepharospasm is. At this visit, participants will receive one of three types of cream. One cream will have a low dose of AH-8, one will have a higher dose of AH-8, and the other will be a placebo (no AH-8).
* One month later, participants will have a followup visit, with tests similar to the first visit. They will also receive more of the cream.
* One month later, participants will have another visit with the same tests. They will be videotaped at this visit to study their facial movements. Those who have responded to the treatment will continue to use the cream. Those who have not responded will be offered the chance to have BoNT injections, and will stop taking the cream.
* One month later, participants who had BoNT injections will have a final visit to check for possible side effects. Those who continued to take the cream will continue on the study.
* The fifth and sixth visits will involve the same tests as before. At the seventh visit, remaining participants will be offered the chance to have BoNT injections, and will stop taking the cream.
* The final visit will check for any side effects from the cream or the injections.

DETAILED DESCRIPTION:
OBJECTIVE:

Test the efficacy of topical AH-8 in blepharospasm treatment.

DESIGN:

This is a randomized, double blind, placebo-controlled study, phase II single center clinical trial. Patients with primary blepharospasm at least 4 months off BoNT therapy with no benefit from last BoNT injection by history and self assesment will be included. We will use 3 study arms placebo and 2 different doses (as concentrations of the AH-8 active substance in the topical preparation). An extension phase is planned after the initial phase.

The patients will have a baseline screening visit, including measurement of the outcome variables, then begin the study intervention. They will have 2 subsequent visits at month 1 and month 2. After this visit, the patients who do not have significant benefit and wish to have an alternative therapy (GROUP 1) will receive BoNT injections according to best practice standards. These patients will then be assessed 1 month later (peak effect of BoNT therapy) and the effect will be compared with the AH-8 effect. The patients who have significant benefit (GROUP 2) will continue therapy for another 4 months (total of 6 months), and will have another assessment at that point. Afterwards the patients will be offered BoNT injections according to best practice standards, similar to Group 1 above, and another assessment will be made one month later (month 7) to compare the effects with AH-8 effects.

OUTCOME MEASURES:

Primary outcome variable: the Jankovic Blepharospasm Rating Scale at month 2.

Secondary outcome variables:

* the Jankovic Blepharospasm Rating Scale at month 1
* the Blepharospasm Disability Scale at month 1
* the Blepharospasm Disability Scale at month 2
* the difference in JBRS at month 3 time point (after BoNT injection) in patients receiving BoNT
* JBRS score at 6 months for patients not receiving BoNT at month 2 (Group 2)
* the difference in JBRS between month 6 and month 7 time point (after BoNT injection) in Group 2 patients
* Blink reflex measures at month 2

Non-parametric comparison (Wilcoxon Mann-Whitney test) of the primary and secondary variables before and after the intervention will be used for statistical analysis. Additional multivariate analysis will explore the influence of other factors (age, gender, disease duration).

Interventions and Duration

Twice daily application of active substance or placebo. Two active substance concentrations, 0.025% and 0.05% AH-8 will be used.

Each subject will be in the study a total of at least 3 months, followed by additional up to 4 months in the second phase for the group 2 patients.

Sample Size and Population

There will be 8 patients per arm, for a total study population of 24. The power calculation for a power of 80%, for a 2-tailed alpha of 0.05, to be able to detect a change of 2 points on the JBRS requires 8 patients per arm. This calculation was based on independent calculation for each dose of the active agent against placebo.

The subjects included will be patients with primary blepharospasm, not currently treated with BoNT (de novo diagnosed patients), but who subjectively express a wish for treatment intervention, with at least one year history from symptom onset, without perceived active change in symptoms by history. Patients with blepharospasm as part of a generalized dystonia or due to a different neurologic condition will be excluded.

Randomization and blinding to be performed by the NIH research pharmacy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Primary blepharospasm diagnosed or confirmed by a Movement Disorders Neurologist, confirmed at the initial visit by a study investigator.
* Individuals off BoNT therapy for at least 4 months will be eligible for this study.

  * Severity prompting need for treatment as determined by clinical judgment
  * At least a score of 4 on the JBRS
  * At least a score of 8 on the BDS
  * Duration of symptoms of at least 1 year, without subjective active progression by patient report
  * Concomitant therapy allowed, except injectable BoNT therapy, provided the doses remain stable throughout the study period
  * Adult patients (> 18)

EXCLUSION CRITERIA:

* Blepharospasm associated with generalized or extensive regional dystonia
* Medical condition impairing the patient's ability to comply with the study protocol or to perform daily applications of the cream as instructed as judged by recruiting physician
* Local eyelid pathology precluding topical treatment
* Received BoNT within 4 months prior to enrollment
* Continued benefit from a prior BoNT injection (by history and self assesment) Current use of cosmetic wrinkle creams
* Prior myectomy procedure excluded
* Pregnant women excluded. Barrier contraception will be used throughout the study for women of childbearing age, as it is not known how the use of hormonal contraceptives may interact with the study substance. Menopausal status will be determined by the CNS IRB criteria. In women of childbearing potential, a pregnancy test will be performed at the initial visit and periodically every 2 months for the duration of the study. Barrier contraception will be deemed necessary for the duration of the study and none after.
* Use of other treatments for blepharospasm allowed if the doses remain constant
* Allergy/sensitivity to study substance or vehicle.
* Active drug or alcohol abuse or dependence
* Patients with uncontrolled co-existing medical conditions: uncontrolled systemic hypertension with values above 170/100; active heart disease needing immediate intervention; active respiratory disease needing intervention; known or observed eye pathology; any condition that would render the patient unable to safely cooperate with the study tests as judged by the screening physician
* Cognitive inability to independently use cr(SqrRoot)(Registered Trademark)me use safely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Codrin I Lungu, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ben Simon GJ, McCann JD. Benign essential blepharospasm. Int Ophthalmol Clin. 2005 Summer;45(3):49-75. doi: 10.1097/01.iio.0000167238.26526.a8. No abstract available. PMID 15970766
- [Background] Defazio G, Livrea P. Primary blepharospasm: diagnosis and management. Drugs. 2004;64(3):237-44. doi: 10.2165/00003495-200464030-00002. PMID 14871168
- [Background] Defazio G, Livrea P. Epidemiology of primary blepharospasm. Mov Disord. 2002 Jan;17(1):7-12. doi: 10.1002/mds.1275. PMID 11835433

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.05% AH-8: Participants in the 0.05% AH-8 arm received the higher dose of the study drug, Acetyl Hexapeptide 8 (AH-8), which is sold under the band name, Argireline.
- 0.025% AH-8: Participants in the 0.025% AH-8 arm received the lower dose of the study drug, Acetyl Hexapeptide 8 (AH-8), which is sold under the band name, Argireline.
Period: Overall Study
Arm/Group | 0.05% AH-8 | 0.025% AH-8 | Placebo
Started | 3 | 2 | 3
Completed | 2 | 2 | 3
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.05% AH-8 | 0.025% AH-8 | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 5
  >=65 years | 1 | 0 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 6
  Male | 2 | 0 | 0 | 2
Jankovic Blepharospasm Rating Scale [Mean (Full Range); unit: units on a scale] — The Jankovic Blepharospasm Rating Scale (JBRS) is a clinical scale measuring the severity and frequency of blepharospasm. Severity and frequency are rated on a 5-point scales ranging from 0 to 4, where 0 indicates no symptoms and 4 indicates the most severe or frequent symptoms. A total score is obtained by adding the severity and frequency subscale scores with total scores ranging from 0 to 8.
  units on a scale | 7 [6 to 8] | 6 [6 to 6] | 6 [5 to 7] | 6.375 [5 to 8]
Blepharospasm Disability Scale [Mean (Full Range); unit: units on a scale] — The Blepharospasm Disability Scale (BDS) is a scale which measures the impact of blepharospasm on the activities of daily living, i.e., need to wear sunglasses (1 or 2) and the impact on the following activities: driving (1 to 5), reading (1 to 3), watching tv (1 to 3), watching movies (1 to 3), shopping (1 to 3), walking about (1 to 4) and housework or job (1 to 3). Patients self-report disability in all areas for a total score between 0 to 26, where 0 indicates no symptoms and 26 indicates severe disability.
  units on a scale | 18 [16 to 21] | 16 [15 to 17] | 17.33 [16 to 19] | 17.25 [15 to 21]

OUTCOME MEASURES:

1. Primary Outcome: The Jankovic Blepharospasm Rating Scale at 2 Month
Description: The Jankovic Blepharospasm Rating Scale (JBRS) at 2 months from the start of the study drug or placebo. The JBRS is a clinical scale measuring the severity and frequency of blepharospasm. Severity and frequency are rated on a 5-point scales ranging from 0 to 4, where 0 indicates no symptoms and 4 indicates the most severe or frequent symptoms (Severity: severe, incapacitating spasm of eyelids and possibly other facial muscles; Frequency: Functionally "blind" due to persistent eye closure (blepharospasm) more than 50% of the waking time.) A total score is obtained by adding the severity and frequency subscale scores with total scores ranging from 0 to 8.
Time Frame: 2 months
Population: One participant in the 0.05% AH-8 arm was withdrawn due to development of blepharitis.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | 0.05% AH-8 | 0.025% AH-8 | Placebo
Number analyzed (Participants) | 2 | 2 | 3
units on a scale | 6 [6 to 6] | 7 [6 to 8] | 4.33 [2 to 6]

2. Secondary Outcome: The Jankovic Blepharospasm Rating Scale at 1 Month
Description: The Jankovic Blepharospasm Rating Scale (JBRS) was measured at 1 month from the start of the study drug or placebo. The JBRS is a clinical scale measuring the severity and frequency of blepharospasm. Severity and frequency are rated on a 5-point scales ranging from 0 to 4, where 0 indicates no symptoms and 4 indicates the most severe or frequent symptoms (Severity: severe, incapacitating spasm of eyelids and possibly other facial muscles; Frequency: Functionally "blind" due to persistent eye closure (blepharospasm) more than 50% of the waking time.) A total score is obtained by adding the severity and frequency subscale scores with total scores ranging from 0 to 8.
Time Frame: 1 month
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | 0.05% AH-8 | 0.025% AH-8 | Placebo
Number analyzed (Participants) | 3 | 2 | 3
units on a scale | 6.66 [6 to 8] | 5.5 [4 to 7] | 5 [2 to 7]

3. Secondary Outcome: The Blepharospasm Disability Scale at 1 Month
Description: The Blepharospasm Disability Scale (BDS) was measured at 1 month from the start of the study drug or placebo. The BDS is a scale which measures the impact of blepharospasm on the activities of daily living, i.e., need to wear sunglasses (1 or 2) and the impact on the following activities: driving (1 to 5), reading (1 to 3), watching tv (1 to 3), watching movies (1 to 3), shopping (1 to 3), walking about (1 to 4) and housework or job (1 to 3). Patients self-report disability in all areas for a total score between 0 to 26, where 0 indicates no symptoms and 26 indicates severe disability.
Time Frame: 1 month
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | 0.05% AH-8 | 0.025% AH-8 | Placebo
Number analyzed (Participants) | 3 | 2 | 3
units on a scale | 16.33 [14 to 20] | 16.5 [16 to 17] | 14.66 [10 to 18]

4. Secondary Outcome: The Blepharospasm Disability Scale at 2 Months
Description: The Blepharospasm Disability Scale (BDS) was measured at 2 months from the start of the study drug or placebo. The BDS is a scale which measures the impact of blepharospasm on the activities of daily living, i.e., need to wear sunglasses (1 or 2) and the impact on the following activities: driving (1 to 5), reading (1 to 3), watching tv (1 to 3), watching movies (1 to 3), shopping (1 to 3), walking about (1 to 4) and housework or job (1 to 3). Patients self-report disability in all areas for a total score between 0 to 26, where 0 indicates no symptoms and 26 indicates severe disability.
Time Frame: 2 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | 0.05% AH-8 | 0.025% AH-8 | Placebo
Number analyzed (Participants) | 2 | 2 | 3
units on a scale | 18.5 [17 to 20] | 15 [12 to 18] | 13.33 [8 to 16]

5. Secondary Outcome: The Jankovic Blepharospasm Rating Scale at 3 Months
Description: The Jankovic Blepharospasm Rating Scale (JBRS) was measured at 3 months from the start of the study drug or placebo. The JBRS is a clinical scale measuring the severity and frequency of blepharospasm. Severity and frequency are rated on a 5-point scales ranging from 0 to 4, where 0 indicates no symptoms and 4 indicates the most severe or frequent symptoms (Severity: severe, incapacitating spasm of eyelids and possibly other facial muscles; Frequency: Functionally "blind" due to persistent eye closure (blepharospasm) more than 50% of the waking time.) A total score is obtained by adding the severity and frequency subscale scores with total scores ranging from 0 to 8.
Time Frame: 3 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | 0.05% AH-8 | 0.025% AH-8 | Placebo
Number analyzed (Participants) | 2 | 2 | 3
units on a scale | 6.5 [6 to 7] | 3 [2 to 4] | 2.33 [1 to 4]

6. Secondary Outcome: The Jankovic Blepharospasm Rating Scale at 6 Months
Description: The Jankovic Blepharospasm Rating Scale (JBRS) was measured at 6 months from the start of the study drug or placebo. The JBRS is a clinical scale measuring the severity and frequency of blepharospasm. Severity and frequency are rated on a 5-point scales ranging from 0 to 4, where 0 indicates no symptoms and 4 indicates the most severe or frequent symptoms (Severity: severe, incapacitating spasm of eyelids and possibly other facial muscles; Frequency: Functionally "blind" due to persistent eye closure (blepharospasm) more than 50% of the waking time.) A total score is obtained by adding the severity and frequency subscale scores with total scores ranging from 0 to 8.
Time Frame: 6 months
Measure: Number; unit: units on a scale
Arm/Group | 0.05% AH-8 | 0.025% AH-8 | Placebo
Number analyzed (Participants) | 1 | 1 | 1
units on a scale | 8 | 6 | 0

7. Secondary Outcome: The Jankovic Blepharospasm Rating Scale at 7 Months
Description: The Jankovic Blepharospasm Rating Scale (JBRS) was measured at 7 months from the start of the study drug or placebo. The JBRS is a clinical scale measuring the severity and frequency of blepharospasm. Severity and frequency are rated on a 5-point scales ranging from 0 to 4, where 0 indicates no symptoms and 4 indicates the most severe or frequent symptoms (Severity: severe, incapacitating spasm of eyelids and possibly other facial muscles; Frequency: Functionally "blind" due to persistent eye closure (blepharospasm) more than 50% of the waking time.) A total score is obtained by adding the severity and frequency subscale scores with total scores ranging from 0 to 8.
Time Frame: 7 months
Measure: Number; unit: units on a scale
Arm/Group | 0.05% AH-8 | 0.025% AH-8 | Placebo
Number analyzed (Participants) | 1 | 0 | 1
units on a scale | 8 |  | 2

ADVERSE EVENTS:
Groups:
- 0.05% AH-8: Participants in the 0.05% AH-8 arm received the higher dose of the study drug, Acetyl Hexapeptide 8 (AH-8), which is sold under the band name, Argireline.
  Topical acetyl hexapeptide-8
- 0.025% AH-8: Participants in the 0.025% AH-8 arm received the lower dose of the study drug, Acetyl Hexapeptide 8 (AH-8), which is sold under the band name, Argireline.
  Topical acetyl hexapeptide-8
- Placebo: Participants in the Placebo arm received the placebo.
  Topical acetyl hexapeptide-8
Arm/Group | 0.05% AH-8 | 0.025% AH-8 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/2 | 1/3
Other Adverse Events (participants affected / at risk) | 2/3 | 0/2 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.05% AH-8 (N=3) | 0.025% AH-8 (N=2) | Placebo (N=3)
Automobile accident (General disorders) | 1 (1) | 0 (0) | 0 (0) — Subject was the driver involved in automobile accident. Subject was on study medication and reported that worsening of blepharospasm may have contributed to accident.
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.05% AH-8 (N=3) | 0.025% AH-8 (N=2) | Placebo (N=3)
Puffiness of lower eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
High blood pressure due to not taking blood pressure medication (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tingling in bilateral eyelids after cream application (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Expected event
Weakness following botulinum toxin injection (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Expected event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes